CLINICAL TRIAL: NCT01498289
Title: A Randomized Phase II Pilot Study Prospectively Evaluating Treatment for Patients Based on ERCC1(Excision Repair Cross-Complementing 1) for Advanced/Metastatic Esophageal, Gastric or Gastroesophageal Junction (GEJ) Cancer
Brief Title: S1201: Combination Chemo for Patients W/Advanced or Metastatic Esophageal, Gastric, or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1201; S1201 (Other: SWOG); U10CA032102 (NIH); NCI-2012-00096 (Other: CTRP)
Record Dates: First submitted 2011-12-22; First posted 2011-12-23 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer; Gastric Cancer
Keywords: recurrent esophageal cancer; stage IV esophageal cancer; recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the gastroesophageal junction; stage IIIB gastric cancer; stage IIIC gastric cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; adenocarcinoma of the esophagus; adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Folfox protocol; Docetaxel; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): FOLFOX regimen: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: FOLFOX regimen — Given IV. Fluorouracil, oxaliplatin, & leucovorin calcium.
  Arms: Arm I
Drug: docetaxel — 30 mg/m^2, IV over 30 minutes on Day 1,8 of each 21 day cycle.
  Other Names: Taxotere; RP56976; NSC-628503
  Arms: Arm II
Drug: fluorouracil — 400 mg/m^2, IV bolus on Day 1 of each 14 day cycle; 2400 mg/m^2 IV over 46-48 hours on Days 1-2 of each 14 day cycle.
  Other Names: 5-fluorouracil; 5-FU; NSC-19893
  Arms: Arm I
Drug: irinotecan hydrochloride — 65 mg/m^2, IV over 90 minutes on Days 1 & 8 of every 21 day cycle.
  Other Names: CPT-11; NSC-616348
  Arms: Arm II
Drug: leucovorin calcium — 400 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
  Other Names: NSC-3590
  Arms: Arm I
Drug: oxaliplatin — 85 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
  Other Names: Eloxatin; NSC-266046
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, fluorouracil, irinotecan hydrochloride, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective in treating tumor cells.

PURPOSE: This randomized phase II trial studies how well oxaliplatin, leucovorin calcium, and fluorouracil work compared to irinotecan hydrochloride and docetaxel in treating patients with esophageal cancer, gastric cancer, or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess progression-free survival of high-excision repair cross-complementing 1(ERCC1) patients with advanced or metastatic cancer of the esophagus, stomach, or gastroesophageal junction (GEJ) treated with FOLFOX comprising oxaliplatin, leucovorin calcium, and fluorouracil compared to those treated with irinotecan hydrochloride plus docetaxel.
* To assess progression-free survival of low-ERCC1 patients with advanced or metastatic cancer of the esophagus, stomach, or GEJ treated with FOLFOX compared to those treated with irinotecan hydrochloride plus docetaxel.
* To assess progression-free survival of low-ERCC1 patients with advanced or metastatic cancer of the esophagus, stomach, or GEJ treated with FOLFOX compared to high-ERCC1 patients treated with FOLFOX.
* To assess overall survival of and toxicities in each of the two treatment arms in this group of patients.
* To assess the response probability (confirmed and unconfirmed, complete and partial responses) in the subset of patients with measurable disease in each of the two treatment arms.
* To explore whether there is evidence of interaction between treatment arm and ERCC1 expression in this group of patients. (Exploratory)
* To bank tissue and blood for future translational medicine studies; a) To explore the relationship of ERCC-1 and ERCC-2 single nucleotide polymorphism (SNP) genotypes with clinical outcome in these patients; and b) To explore the association between germline variations in these SNPs and ERCC-1 mRNA expression in these patients. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to ERCC1 expression (high [≥ 1.7] vs low [< 1.7]), and disease site (esophageal vs gastric/gastroesophageal junction). Patients are randomized to 1 of 2 treatment arms.

* Arm I (FOLFOX): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples may be collected for ERCC1 expression analysis and future research studies.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have unresectable advanced or metastatic histologically or cytologically confirmed adenocarcinoma of the esophagus, stomach, or gastroesophageal junction (GEJ)

  * Patients must not have received treatment for metastatic or unresectable disease
  * Patients must not have brain metastases
* Patients must have measurable and/or non-measurable disease
* Patients who have had HER-2 expression testing prior to patient consent to this study must be HER-2 negative; if HER-2 expression has not been tested prior to patient consent to this study, a second specimen must be submitted for HER-2 expression; if the specimen is HER-2 positive (or if HER-2 could not be evaluated), the patient will not be randomized
* Patients must have completed any prior neoadjuvant and adjuvant therapy for resectable disease at least 180 days prior to registration

PATIENT CHARACTERISTICS:

* Zubrod performance status of 0-1
* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 mg/dL regardless of whether patients have liver involvement secondary to tumor
* AST and ALT both ≤ 3 times institutional upper limit of normal (IULN) unless the liver is involved with tumor, in which case both AST and ALT must be ≤ 5 times IULN
* Serum creatinine < 1.5 mg/dL within 28 days prior to registration AND/OR calculated creatinine clearance > 60 mL/min
* Patients must not have motor or sensory neuropathy > Grade 1 using CTCAE version 4.0
* Patients must not be pregnant or nursing; women and men of reproductive potential must have agreed to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* All palliative radiation therapy alone must be completed at least 14 days prior to registration
* Patient must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other type of therapy for treatment of cancer while on this protocol treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, MD, Principal Investigator — University of Southern California
Locations (508):
- United States (508):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Davis Hospital, Davis, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California at Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Atlo Medical Foundation-Sunnyvale, Sunnyvale, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Breast Cancer Care Consultants, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meredian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Central Illinois CCOP, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants Limited, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Center-West, Kansas City, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center-Shawnee Mission, Shawnee Mission, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology Hematology Associates, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Arnot Ogden Medical Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - New York University Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology and Hematology Care Inc-Taft, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Oncology Inc, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-Charleston, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute/Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Auburn Regional Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Good Samaritan Community Hospital, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 213 participants were randomized, but six were ineligible and 5 were excluded from analysis due to death or withdrawal prior to randomization. Therefore 202 were deemed eligible and analyzable for the primary analysis.
Groups:
- Arm I: FOLFOX regimen: participants receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  FOLFOX regimen: Given IV. Fluorouracil, oxaliplatin, & leucovorin calcium.
  fluorouracil: 400 mg/m^2, IV bolus on Day 1 of each 14 day cycle; 2400 mg/m^2 IV over 46-48 hours on Days 1-2 of each 14 day cycle.
  leucovorin calcium: 400 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
  oxaliplatin: 85 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
- Arm II: IT regimen: participants receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  docetaxel: 30 mg/m^2, IV over 30 minutes on Day 1,8 of each 21 day cycle.
  irinotecan hydrochloride: 65 mg/m^2, IV over 90 minutes on Days 1 & 8 of every 21 day cycle.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 98 | 104
Participants Assessed for AEs | 91 | 98
Completed | 0 | 0
Not Completed | 98 | 104
Not completed — Adverse Event | 16 | 18
Not completed — Death | 6 | 8
Not completed — Withdrawal unrelated to AE | 16 | 16
Not completed — Progression/relapse | 53 | 59
Not completed — Not protocol specified | 7 | 2
Not completed — Reason under review | 0 | 1

BASELINE CHARACTERISTICS:
Population: 213 participants were randomized, but six were ineligible and 5 were excluded from analysis due to death or withdrawal prior to randomization. Therefore 202 were deemed eligible and analyzable for the primary analysis.
Groups:
- Arm II: Participants receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  docetaxel: 30 mg/m^2, IV over 30 minutes on Day 1,8 of each 21 day cycle.
  irinotecan hydrochloride: 65 mg/m^2, IV over 90 minutes on Days 1 & 8 of every 21 day cycle.
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 98 | 104 | 202
Age, Continuous [Median (Full Range); unit: years] | 62.5 [21.5 to 85.6] | 62.4 [33.7 to 84.8] | 62.5 [21.5 to 85.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 78 | 83 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 19 | 31
  Not Hispanic or Latino | 83 | 83 | 166
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 83 | 80 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 10 | 12
ERCC1 [Count of Participants; unit: Participants]
  High (>=1.7) | 13 | 15 | 28
  Low (<1.7) | 85 | 89 | 174
Site of Disease [Count of Participants; unit: Participants]
  Esophageal | 33 | 36 | 69
  Gastric/GEJ | 65 | 68 | 133

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in High-ERCC1 Patients
Description: Progression-free survival is the length of time between protocol registration and disease progression or death, whichever occurs first.
Time Frame: Up to 3 years after registration
Population: Eligible and analyzable participants with ERCC1 level >= 1.7
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I FOLFOX: FOLFOX regimen: Participants receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  FOLFOX regimen: Given IV. Fluorouracil, oxaliplatin, & leucovorin calcium.
  fluorouracil: 400 mg/m^2, IV bolus on Day 1 of each 14 day cycle; 2400 mg/m^2 IV over 46-48 hours on Days 1-2 of each 14 day cycle.
  leucovorin calcium: 400 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
  oxaliplatin: 85 mg/m^2, IV over 2 hours on Day 1 of every 14 day cycle.
- Arm II IT: IT regimen: Participants receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  docetaxel: 30 mg/m^2, IV over 30 minutes on Day 1,8 of each 21 day cycle.
  irinotecan hydrochloride: 65 mg/m^2, IV over 90 minutes on Days 1 & 8 of every 21 day cycle.
Arm/Group | Arm I FOLFOX | Arm II IT
Number analyzed (Participants) | 13 | 15
months | 4.7 [2.1 to 8.7] | 5.3 [0.9 to 11.5]
Statistical Analysis 1: Comparison: Arm I FOLFOX vs Arm II IT; Test type: Superiority; p = 0.83, Regression, Cox; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.41 to 2.05]

2. Primary Outcome: PFS in Low-ERCC1 Participants
Description: as for outcome 1
Time Frame: Up to 3 years after registration
Population: Eligible and analyzable participants with ERCC1 level < 1.7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 85 | 89
months | 5.9 [4.1 to 7.1] | 2.8 [1.7 to 4.1]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.50 to 0.93]

3. Primary Outcome: Overall Survival (OS)
Description: OS is the length of time between protocol registration and patient death
Time Frame: Up to 3 years after registration
Population: Eligible and analyzable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 98 | 104
months | 11.4 [9.8 to 13.5] | 8.7 [6.0 to 10.1]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.20, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.61 to 1.11]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR (complete response, unconfirmed complete response, partial response, unconfirmed partial response) in patients with measurable disease were assessed in each arm and compared between arms using Chi-squared test.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years after registration
Population: Participants with measurable disease
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 79 | 88
percentage of evaluable participants | 42 [31 to 53] | 30 [20 to 39]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.10, Chi-squared

5. Secondary Outcome: PFS Variation by ERCC1
Description: Progression-free survival is the length of time between protocol registration and disease progression or death, whichever occurs first.
  Participants were divided into subgroups according to ERCC1 quartiles to assess whether the differences in PFS between the two treatment arms varied by ERCC1 levels.
Time Frame: up to 3 years after registration
Population: Eligible and analyzable participants were divided into quartiles based on ERCC1 levels.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 98 | 104
months
  Q1 ERCC1 (0.20-0.80): number analyzed (Participants) | 24 | 26
  Q1 ERCC1 (0.20-0.80) | 5.6 [2.4 to 8.3] | 2.8 [1.4 to 4.9]
  Q2 ERCC1 (0.81-1.10): number analyzed (Participants) | 25 | 26
  Q2 ERCC1 (0.81-1.10) | 7.4 [4.1 to 9.1] | 3.0 [1.9 to 4.2]
  Q3 ERCC1 (1.11-1.42): number analyzed (Participants) | 27 | 23
  Q3 ERCC1 (1.11-1.42) | 5.6 [2.9 to 7.0] | 2.9 [1.0 to 4.7]
  Q4 ERCC1 (1.43-5.71): number analyzed (Participants) | 22 | 29
  Q4 ERCC1 (1.43-5.71) | 4.6 [2.1 to 8.7] | 2.6 [1.3 to 5.6]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Statistical analysis for Q1 ERCC1; Test type: Superiority; p = 0.41, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.44 to 1.40]
Statistical Analysis 2: Comparison: Arm I vs Arm II; Statistical analysis for Q2 ERCC1; Test type: Superiority; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.32 to 1.02]
Statistical Analysis 3: Comparison: Arm I vs Arm II; Statistical analysis for Q3 ERCC1; Test type: Superiority; p = 0.66, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.49 to 1.58]
Statistical Analysis 4: Comparison: Arm I vs Arm II; Statistical analysis for Q4 ERCC1; Test type: Superiority; p = 0.30, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.42 to 1.31]

6. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Participants who received at least one dose of protocol treatment and were thus eligible for AE assessment
Measure: Number; unit: Participants
Groups:
- Arm I FOLFOX: FOLFOX regimen: participants receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. FOLFOX regimen: Given IV. Fluorouracil, oxaliplatin, and leucovorin calcium.
- Arm II IT: IT regimen: participants receive irinotecan hydrochloride IV over 90 minutes and docetaxel IV over 30-60 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. docetaxel: 30 mg/m^2, IV over 30 minutes on Day 1,8 of each 21 day cycle.
Arm/Group | Arm I FOLFOX | Arm II IT
Number analyzed (Participants) | 91 | 98
Participants
  Abdominal pain | 1 | 0
  Activated partial thromboplastin time prolonged | 0 | 1
  Acute kidney injury | 0 | 1
  Alanine aminotransferase increased | 2 | 1
  Alkaline phosphatase increased | 1 | 1
  Allergic reaction | 1 | 0
  Anemia | 6 | 14
  Anorexia | 0 | 7
  Aspartate aminotransferase increased | 2 | 5
  Back pain | 0 | 1
  Bladder infection | 0 | 1
  Blood bilirubin increased | 1 | 1
  Bone pain | 1 | 0
  CD4 lymphocytes decreased | 0 | 3
  Confusion | 1 | 0
  Death NOS | 1 | 0
  Dehydration | 2 | 19
  Depression | 1 | 0
  Diarrhea | 4 | 28
  Dry mouth | 1 | 0
  Dysphagia | 1 | 1
  Edema limbs | 0 | 1
  Esophageal hemorrhage | 0 | 1
  Esophagitis | 0 | 1
  Fatigue | 7 | 14
  Febrile neutropenia | 1 | 6
  Gastrointestinal pain | 0 | 1
  Generalized muscle weakness | 2 | 2
  Headache | 0 | 1
  Heart failure | 0 | 1
  Hyperglycemia | 1 | 1
  Hypertension | 1 | 1
  Hypoalbuminemia | 1 | 4
  Hypocalcemia | 0 | 2
  Hypokalemia | 2 | 8
  Hypomagnesemia | 0 | 2
  Hyponatremia | 2 | 5
  Hypotension | 1 | 3
  INR increased | 0 | 1
  Infections and infestations - Other, specify | 0 | 1
  Infusion related reaction | 1 | 0
  Leukocytosis | 0 | 1
  Lung infection | 1 | 1
  Lymphocyte count decreased | 9 | 7
  Mucositis oral | 2 | 1
  Multi-organ failure | 0 | 2
  Nausea | 7 | 12
  Neutrophil count decreased | 29 | 19
  Non-cardiac chest pain | 0 | 1
  Obstruction gastric | 1 | 0
  Palmar-plantar erythrodysesthesia syndrome | 1 | 0
  Peripheral motor neuropathy | 1 | 0
  Peripheral sensory neuropathy | 10 | 1
  Platelet count decreased | 5 | 1
  Pneumonitis | 0 | 1
  Respiratory failure | 0 | 2
  Sepsis | 1 | 6
  Stomach pain | 0 | 2
  Syncope | 1 | 2
  Thromboembolic event | 1 | 0
  Upper gastrointestinal hemorrhage | 0 | 1
  Urinary tract infection | 0 | 1
  Vascular access complication | 0 | 1
  Vomiting | 5 | 8
  Weight loss | 0 | 2
  White blood cell decreased | 9 | 14

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Population description for all-cause mortality: all eligible and analyzable participants
  Population description for AEs: participants who received at least one dose of protocol treatment and were thus assessed for AEs
Arm/Group | Arm I FOLFOX | Arm II IT
All-Cause Mortality (participants affected / at risk) | 89/98 | 94/104
Serious Adverse Events (participants affected / at risk) | 7/91 | 17/98
Other Adverse Events (participants affected / at risk) | 88/91 | 95/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I FOLFOX (N=91) | Arm II IT (N=98)
Diarrhea (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 2 | 4
Multi-organ failure (General disorders) | 0 | 2
Sudden death NOS (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 6
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I FOLFOX (N=91) | Arm II IT (N=98)
Anemia (Blood and lymphatic system disorders) | 65 | 70
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorders-Other (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 9
Hearing impaired (Ear and labyrinth disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Endocrine disorders-Other (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 6 | 4
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 3
Eye disorders-Other (Eye disorders) | 0 | 3
Eye pain (Eye disorders) | 2 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 32 | 40
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 5 | 4
Bloating (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 43 | 33
Diarrhea (Gastrointestinal disorders) | 33 | 68
Dry mouth (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 7
Dysphagia (Gastrointestinal disorders) | 25 | 23
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 1
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 3 | 4
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 6
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 7 | 8
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 4
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 3 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 4 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Jejunal stenosis (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 30 | 9
Nausea (Gastrointestinal disorders) | 60 | 62
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 2 | 4
Toothache (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 38 | 44
Chills (General disorders) | 9 | 5
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 20 | 25
Edema trunk (General disorders) | 0 | 1
Facial pain (General disorders) | 3 | 0
Fatigue (General disorders) | 74 | 71
Fever (General disorders) | 6 | 12
Flu like symptoms (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 1
General disorders and admin site conditions - Other (General disorders) | 3 | 0
Infusion related reaction (General disorders) | 2 | 2
Injection site reaction (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 5 | 6
Pain (General disorders) | 8 | 6
Gallbladder pain (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 6 | 3
Bladder infection (Infections and infestations) | 0 | 2
Bronchial infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 2 | 4
Lip infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Lymph gland infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 2
Otitis media (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Rhinitis infective (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 3 | 4
Tooth infection (Infections and infestations) | 0 | 3
Tracheitis (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 3 | 0
Burn (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 19 | 20
Alkaline phosphatase increased (Investigations) | 39 | 31
Aspartate aminotransferase increased (Investigations) | 26 | 28
Blood bilirubin increased (Investigations) | 13 | 10
CD4 lymphocytes decreased (Investigations) | 4 | 7
Cholesterol high (Investigations) | 2 | 2
Creatinine increased (Investigations) | 2 | 13
Ejection fraction decreased (Investigations) | 0 | 1
INR increased (Investigations) | 1 | 3
Investigations-Other (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 27 | 26
Neutrophil count decreased (Investigations) | 47 | 30
Platelet count decreased (Investigations) | 50 | 12
Serum amylase increased (Investigations) | 0 | 1
Weight gain (Investigations) | 5 | 2
Weight loss (Investigations) | 37 | 32
White blood cell decreased (Investigations) | 50 | 41
Anorexia (Metabolism and nutrition disorders) | 40 | 46
Dehydration (Metabolism and nutrition disorders) | 13 | 35
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 42 | 36
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 44 | 51
Hypocalcemia (Metabolism and nutrition disorders) | 30 | 34
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 4
Hypokalemia (Metabolism and nutrition disorders) | 20 | 31
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 9
Hyponatremia (Metabolism and nutrition disorders) | 21 | 35
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 | 17
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 6
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 16 | 20
Dysesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 19 | 19
Dysphasia (Nervous system disorders) | 1 | 2
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 11 | 9
Hypersomnia (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Nervous system disorders-Other (Nervous system disorders) | 3 | 0
Paresthesia (Nervous system disorders) | 18 | 3
Peripheral motor neuropathy (Nervous system disorders) | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 57 | 18
Sinus pain (Nervous system disorders) | 0 | 2
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 4
Tremor (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 15 | 16
Confusion (Psychiatric disorders) | 3 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 15 | 9
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 14 | 13
Libido decreased (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Psychiatric disorders-Other (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Chronic kidney disease (Renal and urinary disorders) | 2 | 3
Hematuria (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 3
Urinary retention (Renal and urinary disorders) | 2 | 2
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Nipple deformity (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 4
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 5 | 2
Hypertension (Vascular disorders) | 18 | 15
Hypotension (Vascular disorders) | 7 | 19
Thromboembolic event (Vascular disorders) | 10 | 7
Vascular disorders-Other (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-04-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT01498289/Prot_SAP_ICF_000.pdf